CLINICAL TRIAL: NCT04502472
Title: Treatment of Severe Coronavirus Disease 2019 (COVID-19) With Convalescent Plasma Collected From Individuals With Documented Infection and Recovery From COVID-19 (SARS-CoV-2)
Brief Title: Treatment of Severe Coronavirus Disease 2019 (COVID-19) With Convalescent Plasma
Acronym: Inova-CCP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: FDA gave emergency use approval to COVID-19 convalescent plasma on 08/24/2020
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inova COVID-19 CCP
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase 1 will be recruitment and enrollment of plasma donors. Phase 2 will be continued recruitment and enrollment of plasma donors, with the addition of recruitment and enrollment of plasma recipients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion (Experimental): Patients hospitalized with COVID-19 infection with severe or life-threatening clinical syndrome and meet eligibility criteria
  Interventions: Biological: Convalescent plasma transfusion

INTERVENTIONS:
Biological: Convalescent plasma transfusion — Transfusion of COVID-19 convalescent plasma to participants currently hospitalized with COVID-19 infection with severe or life-threatening clinical syndrome.

SUMMARY:
The investigators hypothesize that use of convalescent plasma donated from individuals recovered from Coronavirus Disease 2019 (COVID-19) will help expedite recovery of individuals with active, severe COVID-19 infection.

DETAILED DESCRIPTION:
The purpose of this research study is to see if convalescent plasma is safe and effective for the treatment of patients acutely ill with COVID-19. The researchers want to confirm the right dose levels of immunoglobulins/antibodies (immune proteins) and find out what therapeutic effects plasma donated by recovered individuals has on people severely sick with COVID-19.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

Inclusion Criteria for Convalescent Plasma Donors:

- Outpatients 18 years old and older who have recovered from COVID-19:

* Have proof of Original Positive SARS-CoV-2 NAT nasopharyngeal (NP) test result
* Complete resolution of symptoms at least 14 days prior to donation
* Negative SARS-CoV-2 NAT nasopharyngeal (NP) specimen at screening visit
* Able to meet standard criteria for blood donation
* Clinically stable based on provider assessment

Phase 1 Exclusion Criteria:

Exclusion criteria:

* Inability to complete or contraindication to donation based on Donor History -
* Questionnaire (DHQ), FDA approved standard blood donation form
* Hb<13.0 g/dL for males
* Hb<12.5 g/dL for females
* History of 3 more pregnancies unless HLA antibody testing is performed and deemed acceptable by director of blood donor services (to reduce risks of transfusion Related Acute Lung Injury in recipients). The presence of any transfusion transmitted diseases is based on history or test results from blood sample collected from the donor at time of plasma collection in accordance to standard practice.
* Female subjects who are pregnant by self-report.
* Receipt of pooled immunoglobulin in past 30 days

PHASE 2: Inclusion Criteria for Recipients of COVID-19 Convalescent Plasma:

* Patients in the Inova Health System with confirmed COVID-19 by PCR testing
* Age ≥ 13 years
* Currently hospitalized with COVID-19 infection with severe or life-threatening clinical syndrome as follows:
* Severe COVID-19: (three or more of the following)

  * Dyspnea
  * Respiratory rate ≥ 30/min
  * Blood oxygen saturation (SpO2) ≤ 94% on room air
  * Partial pressure of arterial oxygen to fraction of inspired oxygen (P:F) ratio < 300
  * Pulmonary infiltrates > 50% of lung parenchyma within 24 to 48 hours
* Life-threatening disease is defined as: (one of the following)

  * Respiratory failure
  * Septic shock, and/or
  * Multiple organ dysfunction or failure
* Patient must provide informed consent or have health care power of attorney/next of kin provide consent if he/she cannot.

PHASE 2 Exclusion Criteria:

* Contraindication to receive plasma as deemed by the treating physician
* Severe hypercoagulable state (documented in medical chart or by treating physician assessment)
* Absolute IgA deficiency
* Prior history of Transfusion Related Acute Lung Injury (TRALI)
* Inability to tolerate plasma volume due to severe systolic or diastolic heart failure despite slower infusion and diuretic administration
* Positive pregnancy test (HCG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Brown, M.D., Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marano G, Vaglio S, Pupella S, Facco G, Catalano L, Liumbruno GM, Grazzini G. Convalescent plasma: new evidence for an old therapeutic tool? Blood Transfus. 2016 Mar;14(2):152-7. doi: 10.2450/2015.0131-15. Epub 2015 Nov 6. PMID 26674811
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Maiztegui JI, Fernandez NJ, de Damilano AJ. Efficacy of immune plasma in treatment of Argentine haemorrhagic fever and association between treatment and a late neurological syndrome. Lancet. 1979 Dec 8;2(8154):1216-7. doi: 10.1016/s0140-6736(79)92335-3. PMID 92624
- [Background] Soo YO, Cheng Y, Wong R, Hui DS, Lee CK, Tsang KK, Ng MH, Chan P, Cheng G, Sung JJ. Retrospective comparison of convalescent plasma with continuing high-dose methylprednisolone treatment in SARS patients. Clin Microbiol Infect. 2004 Jul;10(7):676-8. doi: 10.1111/j.1469-0691.2004.00956.x. PMID 15214887
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Background] van Griensven J, Edwards T, Baize S; Ebola-Tx Consortium. Efficacy of Convalescent Plasma in Relation to Dose of Ebola Virus Antibodies. N Engl J Med. 2016 Dec 8;375(23):2307-2309. doi: 10.1056/NEJMc1609116. Epub 2016 Nov 14. No abstract available. PMID 27959686
- [Background] WHO. Use of convalescent whole blood or plasma collected from patients recovered from Ebola virus disease for transfusion, as an empirical treatment during outbreaks. 2014 http://apps.who.int/iris/rest/bitstreams/604045/retrieve (accessed 3/27/2020).
- [Background] WHO. Clinical management of severe acute respiratory infection when novel coronavirus (nCoV) infection is suspected 2020. https://www.who.int/docs/default-source/coronaviruse/clinical-management-of-novel-cov.pdf (accessed 3/27/20).
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Background] Amanat F, Stadlbauer D, Strohmeier S, Nguyen THO, Chromikova V, McMahon M, Jiang K, Arunkumar GA, Jurczyszak D, Polanco J, Bermudez-Gonzalez M, Kleiner G, Aydillo T, Miorin L, Fierer DS, Lugo LA, Kojic EM, Stoever J, Liu STH, Cunningham-Rundles C, Felgner PL, Moran T, Garcia-Sastre A, Caplivski D, Cheng AC, Kedzierska K, Vapalahti O, Hepojoki JM, Simon V, Krammer F. A serological assay to detect SARS-CoV-2 seroconversion in humans. Nat Med. 2020 Jul;26(7):1033-1036. doi: 10.1038/s41591-020-0913-5. Epub 2020 May 12. PMID 32398876
- [Background] Epstein J, Burnouf T. Points to consider in the preparation and transfusion of COVID-19 convalescent plasma. Vox Sang. 2020 Aug;115(6):485-487. doi: 10.1111/vox.12939. Epub 2020 May 14. No abstract available. PMID 32319102
- [Background] Beigel JH, Tebas P, Elie-Turenne MC, Bajwa E, Bell TE, Cairns CB, Shoham S, Deville JG, Feucht E, Feinberg J, Luke T, Raviprakash K, Danko J, O'Neil D, Metcalf JA, King K, Burgess TH, Aga E, Lane HC, Hughes MD, Davey RT; IRC002 Study Team. Immune plasma for the treatment of severe influenza: an open-label, multicentre, phase 2 randomised study. Lancet Respir Med. 2017 Jun;5(6):500-511. doi: 10.1016/S2213-2600(17)30174-1. Epub 2017 May 15. PMID 28522352
- [Background] Wang Y, Fan G, Horby P, Hayden F, Li Q, Wu Q, Zou X, Li H, Zhan Q, Wang C, Cao B; CAP-China Network. Comparative Outcomes of Adults Hospitalized With Seasonal Influenza A or B Virus Infection: Application of the 7-Category Ordinal Scale. Open Forum Infect Dis. 2019 Feb 15;6(3):ofz053. doi: 10.1093/ofid/ofz053. eCollection 2019 Mar. PMID 30895200
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Woelfel R, Corman VM, Guggemos W, et al. Clinical presentation and virological assessment of hospitalized cases of coronavirus disease 2019 in a travel-associated transmission cluster. BMJ Yale 2020. https://doi.org/10.1101/2020.03.05.20030502
- [Background] Pandey S, Vyas GN. Adverse effects of plasma transfusion. Transfusion. 2012 May;52 Suppl 1(Suppl 1):65S-79S. doi: 10.1111/j.1537-2995.2012.03663.x. PMID 22578374

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-19 Convalescent Plasma (CCP) Donors: Patients recovered from COVID-19 and donated CCP through the study.
- COVID-19 Convalescent Plasma (CCP Recipients): Patients who were hospitalized with COVID-19 and received CCP infusions through the study.
Period: Overall Study
Arm/Group | COVID-19 Convalescent Plasma (CCP) Donors | COVID-19 Convalescent Plasma (CCP Recipients)
Started | 61 | 48
Completed | 58 | 45
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Donor of COVID-19 Convalescent Plasma (CCP): Patients who recovered from COVID-19 infection and test negative for COVID-19 by nasopharyngeal swab.
- Total: Total of all reporting groups
Arm/Group | Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion | Donor of COVID-19 Convalescent Plasma (CCP) | Total
Number analyzed (Participants) | 48 | 61 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 31 | 54 | 85
  >=65 years | 16 | 7 | 23
Age, Continuous [Mean (Full Range); unit: years] | 59 [16 to 87] | 48 [18 to 80] | 53 [16 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 65
  Male | 18 | 26 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 4 | 31
  Not Hispanic or Latino | 20 | 54 | 74
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 12 | 53 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 3 | 30
Region of Enrollment [Number; unit: participants]
  United States | 48 | 61 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change is Clinical Status
Description: Change is clinical status as captured by 7-point ordinal scale to include
  1. Death
  2. Hospitalized, requiring mechanical ventilation or ECMO
  3. Hospitalized, requiring non-invasive ventilation or high flow oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen--requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen-not requiring ongoing medical care (COVID-19 related or otherwise).
  7. Not Hospitalized
Time Frame: Time of plasma infusion (day 0) compared to day 7
Population: Patients that were hospitalized with COVID-19 and received CCP were evaluated using the 7-point ordinal scale. The worse oxygenation status was used for day 0 and day 7.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Patients Hospitalized With COVID-19: 45 patients were hospitalized with COVID-19 and received CCP through the study.
Arm/Group | Patients Hospitalized With COVID-19
Number analyzed (Participants) | 45
units on a scale
  Average Day 1 Ordinal Scale | 3.06 [1 to 7]
  Average Day 7 Ordinal Scale | 3.86 [1 to 7]

2. Primary Outcome: Transfusion Related Events Due to Administration of CCP
Description: Number of participants with Transfusion Related Adverse Events
Time Frame: Within 6 hours of infusion
Population: Transfusion related events were only measured in the convalescent plasma recipient arm. 48 patients were enrolled in the study. 45 received CCP. 3 patients received CCP through individual INDs.
  This outcome measure was only for patients who were hospitalized with COVID-19 and received CCP through the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Hospitalized With COVID-19
Number analyzed (Participants) | 45
Participants | 3

3. Secondary Outcome: Change is Clinical Status
Description: Change in 7-point ordinal scale score from time of plasma infusion (day 0-prior to first infusion) to days 7, 14, 21, and 28.
  7 point ordinal scale:
  1. Death
  2. Hospitalized, requiring mechanical ventilation or ECMO
  3. Hospitalized, requiring non-invasive ventilation or high flow oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen--requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen-not requiring ongoing medical care (COVID-19 related or otherwise).
  7. Not Hospitalized
Time Frame: Time of plasma infusion (day 0 prior to first infusion) to days 7,14, 21, and 28
Population: Patients ts that were hospitalized with COVID-19 and received CCP were evaluated using the 7-point ordinal scale. The worse oxygenation status was used for days 7, 14, 21, and 28
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Hospitalized With COVID-19
Number analyzed (Participants) | 45
Participants
  Ordinal Scale Day 0: Ordinal Scale 2 out of 7 | 10
  Ordinal Scale Day 0: Ordinal Scale 3 out of 7 | 22
  Ordinal Scale Day 0: Ordinal Scale 4 out of 7 | 13
  Ordinal Scale Day 0: Ordinal Scale 5 out of 7 | 0
  Ordinal Scale Day 0: Ordinal Scale 6 out of 7 | 0
  Ordinal Scale Day 0: Ordinal Scale 7 out of 7 | 0
  Ordinal Scale Day 0: Ordinal Scale 1 out of 7 | 0
  Ordinal Scale Day 7: Ordinal Scale 2 out of 7 | 11
  Ordinal Scale Day 7: Ordinal Scale 3 out of 7 | 6
  Ordinal Scale Day 7: Ordinal Scale 4 out of 7 | 10
  Ordinal Scale Day 7: Ordinal Scale 5 out of 7 | 1
  Ordinal Scale Day 7: Ordinal Scale 6 out of 7 | 0
  Ordinal Scale Day 7: Ordinal Scale 7 out of 7 | 12
  Ordinal Scale Day 7: Ordinal Scale 1 out of 7 | 5
  Ordinal Scale Day 14: Ordinal Scale 2 out of 7 | 5
  Ordinal Scale Day 14: Ordinal Scale 3 out of 7 | 3
  Ordinal Scale Day 14: Ordinal Scale 4 out of 7 | 5
  Ordinal Scale Day 14: Ordinal Scale 5 out of 7 | 0
  Ordinal Scale Day 14: Ordinal Scale 6 out of 7 | 0
  Ordinal Scale Day 14: Ordinal Scale 7 out of 7 | 21
  Ordinal Scale Day 14: Ordinal Scale 1 out of 7 | 11
  Ordinal Scale Day 21: Ordinal Scale 2 out of 7 | 5
  Ordinal Scale Day 21: Ordinal Scale 3 out of 7 | 1
  Ordinal Scale Day 21: Ordinal Scale 4 out of 7 | 3
  Ordinal Scale Day 21: Ordinal Scale 5 out of 7 | 0
  Ordinal Scale Day 21: Ordinal Scale 6 out of 7 | 0
  Ordinal Scale Day 21: Ordinal Scale 7 out of 7 | 23
  Ordinal Scale Day 21: Ordinal Scale 1 out of 7 | 13
  Ordinal Scale Day 28: Ordinal Scale 2 out of 7 | 2
  Ordinal Scale Day 28: Ordinal Scale 3 out of 7 | 2
  Ordinal Scale Day 28: Ordinal Scale 4 out of 7 | 1
  Ordinal Scale Day 28: Ordinal Scale 5 out of 7 | 0
  Ordinal Scale Day 28: Ordinal Scale 6 out of 7 | 0
  Ordinal Scale Day 28: Ordinal Scale 7 out of 7 | 26
  Ordinal Scale Day 28: Ordinal Scale 1 out of 7 | 14

4. Secondary Outcome: Length of Hospital Stay
Description: Total duration of hospital stay which includes from Admission with COVID-19 from admission with COVID-19 symptoms to discharge or death (up to an average of 67 days)
Time Frame: Total Index Hospitalization
Population: Total duration of hospital stay which includes from Admission with COVID-19 from admission with COVID-19 symptoms to discharge or death
Measure: Mean (Full Range); unit: days
Arm/Group | Patients Hospitalized With COVID-19
Number analyzed (Participants) | 45
days | 20 [4 to 67]

5. Secondary Outcome: Mechanical Ventilation
Description: Number of participants that required mechanical ventilation that were not on mechanical ventilation at that time point.
Time Frame: Days 7, 14, 21, 28
Population: The count of participants below shows the total number of participants needing mechanical ventilation for that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion
Number analyzed (Participants) | 45
Participants
  Day 7: Patients requiring mechanical ventilation | 11
  Day 7: Patients not requiring mechanical ventilation | 17
  Day 7: Patients deceased | 5
  Day 7: Patients discharged | 12
  Day 14: Patients requiring mechanical ventilation | 5
  Day 14: Patients not requiring mechanical ventilation | 8
  Day 14: Patients deceased | 11
  Day 14: Patients discharged | 21
  Day 21: Patients requiring mechanical ventilation | 5
  Day 21: Patients not requiring mechanical ventilation | 4
  Day 21: Patients deceased | 13
  Day 21: Patients discharged | 23
  Day 28: Patients requiring mechanical ventilation | 2
  Day 28: Patients not requiring mechanical ventilation | 3
  Day 28: Patients deceased | 14
  Day 28: Patients discharged | 26

6. Secondary Outcome: Change in Mechanical Ventilation Status
Description: Number of participants who required a change in the mechanical ventilation status
Time Frame: Day 0 (date of CCP transfusion) to Day 28
Population: Patients that were hospitalized with COVID-19 and received CCP through the study
Measure: Count of Participants; unit: Participants
Groups:
- Patients Hospitalized With COVID-19: 45 patients were analyzed
Arm/Group | Patients Hospitalized With COVID-19
Number analyzed (Participants) | 45
Participants | 6

7. Secondary Outcome: Mortality
Description: All-cause Mortality
Time Frame: From Day of Transfusion (Day 0) to Day 28 post-transfusion for patients who received CCP. Patients who donated CCP were not followed for a defined time period after CCP donation.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Recovered From COVID-19: patients who donated CCP
Arm/Group | Patients Hospitalized With COVID-19 | Patients Recovered From COVID-19
Number analyzed (Participants) | 45 | 61
Participants | 14 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for up to 67 days
Description: Only serious adverse events were recorded.
Groups:
- Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion: Patients hospitalized with COVID-19 infection with severe or life-threatening clinical syndrome and meet eligibility criteria
  Convalescent plasma transfusion: Transfusion of COVID-19 convalescent plasma to participants currently hospitalized with COVID-19 infection with severe or life-threatening clinical syndrome.
  Adverse Events only monitored/assessed in Convalescent Plasma Recipients.
Arm/Group | Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion
All-Cause Mortality (participants affected / at risk) | 14/45
Serious Adverse Events (participants affected / at risk) | 21/45
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion (N=45)
Death (Respiratory, thoracic and mediastinal disorders) | 14 (14) — 14 patients died during the study.
transfusion reaction (Blood and lymphatic system disorders) | 3 (3) — 3 patients had a transfusion reaction due to CCP.
Intubation (Respiratory, thoracic and mediastinal disorders) | 4 (4) — 4 patients were intubated during the course of the study that recovered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT04502472/Prot_SAP_002.pdf